CLINICAL TRIAL: NCT00910572
Title: Radioembolization With Yttrium-90 Microspheres for Intermediate or Advanced HCC (Hepatocellular Carcinoma) Not Eligible to Curative Approach. A Phase II-b Study.
Brief Title: Radioembolization With Yttrium-90 Microspheres for Intermediate or Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: Gastro Intestinal Surgery and Liver Transplantation (Unknown); The Hepato-Oncology Group: Department of Surgery, Medicine and Radiology (Unknown)
Responsible Party: Dr. Vincenzo Mazzaferro, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INT 30/90
Record Dates: First submitted 2009-05-28; First posted 2009-06-01 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2009-05

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: Yttrium-90; Radiation; Radioembolization; Hepatoma; BCLC classification; Hepatic loco-regional treatments; Yttrium; Microspheres
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Yttrium-90 microspheres (Therasphere MDS Nordion) — Y-90 is incorporated into very tiny glass beads (microspheres: Therasphere MDS Nordion) and is injected into the liver tumor through the hepatic arteries, which are responsible for the feeding of the neoplastic liver tissue. Since the microspheres are unable to pass through the micro-vasculature of the liver parenchyma and tumor they are trapped at those sites and exert a local radio-therapeutic effect.
  Other Names: Therasphere, produced by MDS Nordion, Ottawa, Canada

SUMMARY:
Rationale: Patients diagnosed with hepatocellular carcinoma (HCC) at an intermediate or advanced stage (according to the BCLC classification system) are not amenable of curative treatment. According to EASL and AASLD guidelines patients with an intermediate stage HCC are treated with trans-arterial chemoembolization (TACE) while patients with an advanced stage HCC are treated with molecular targeted drugs or other combinations according to their liver function. The median survival expected for patients in intermediate-advanced stages ranges from 11 to 20 months.

Purpose of the Study: The purpose of this prospective phase II study is to determine whether or not Radioembolization with Yttrium-90 microspheres (TheraSphere®) provides an anti-tumoral effect and a sensible benefit in terms of time-to-progression (TTP) and survival in patients with good liver function (Child A-B7) and a confirmed diagnosis of Intermediate or Advanced (because of the presence of neoplastic portal thrombosis) Hepatocellular Carcinoma (HCC).

DETAILED DESCRIPTION:
Patients at an intermediate stage (BCLC-B) are currently offered trans-arterial chemoembolisation (TACE) as the standard of care. A recent meta-analysis showed that radioembolization with beta-emitting Yttrium-90-loaded glass microspheres (TheraSphere®) in patients with HCC achieves a median objective response in 79% of cases (range 29-88%) and median survival exceeding 15 months has been reported in patients at intermediate stages who have been treated with TheraSphere®.

In patients with HCC at an advanced stage (BCLC-C) the single treatment that has shown a statistical advantage on overall survival and disease progression is sorafenib, that provides a median survival of 10.7 months. Based on the results reported in literature, the estimated median expected survival of patients with advanced HCC treated by TheraSphere® can be as long as 12 months.

After approval on July 2007 of a treatment protocol of Y-90 for compassionate use by the institutional IRB, at the National Cancer Institute of Milan 40 consecutive patients have been treated with radioembolization with Yttrium-90 microspheres (Theraspheres®) according to the same guidelines of the present prospective phase II protocol. The initial series of 40 patients treated according to a compassionate use of Y-90 has been instrumental for the assessment of the procedure's safety and tolerability. The present study has been targeted to 60 cases including the fist series of 40 "compassionate" patients, due to their adherence to the same inclusion/exclusion criteria of the proposed phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of HCC confirmed by histology or non-invasive criteria (EASL/AASLD)
2. Intermediate stage (BCLC-B) HCC: patients with a large or multinodular HCC (single HCC > 5 cm or multiple HCC defined as > 3 nodules > 3 cm), a Child Pugh class A or B7 and no cancer related symptoms (PS=0-1).
3. Advanced stage (BCLC-C) HCC: patients with hepatic vascular involvement (at any tumor number and diameter), a Child Pugh class A or B7, no cancer related symptoms (PS=0-1) and absence of extra-hepatic tumor spread.
4. Cancer-related symptoms within the ECOG 0-1 score
5. Liver function within Child B-7 class
6. Platelets > 50.000/µL
7. WBC > 1500/µL
8. AST/ALT < 5 times the upper limit of normal (U/L)
9. Creatinine < 2.0 mg /dL
10. No indication for any possible curative treatment after multidisciplinary assessment (resection, ablation, transplantation)
11. Signed informed consent

Exclusion Criteria:

1. Child-Pugh class higher than B-7 at entry
2. ECOG performance score ≥ 2 at entry
3. Tumor volume ≥ 50% of liver volume
4. Extrahepatic tumor spread
5. Pulmonary insufficiency
6. Life expectancy of less than 3 months due to HCC or less than 6 months due to any other disease
7. Previous chemoembolization procedure (TACE)
8. Evidence on 99mTc-MAA scan of vascular shunts that can not be corrected by angiographic coil embolization
9. Evidence on 99mTc-MAA scan of lung shunting, with a potential absorbed dose of radiation to the lungs > 30 Gy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Time to progression (TTP) | At 1, 3, 6, 12 months and every 6 months thereafter

SECONDARY OUTCOMES:
Tumor Response according to RECIST, WHO, EASL and Choi criteria | At 3, 6, 12 months and every 6 months thereafter
Overall survival | At 1, 3, 6, 12 months and every 6 months thereafter
Safety: documentation of all adverse events | At 1, 3, 6, 12 months and every 6 months thereafter
Time-to-symptomatic progression (TTSP) | At 1, 3, 6, 12 months and every 6 months thereafter

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Mazzaferro, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milano, Milan, Italy

REFERENCES:
- [Background] Salem R, Lewandowski RJ, Atassi B, Gordon SC, Gates VL, Barakat O, Sergie Z, Wong CY, Thurston KG. Treatment of unresectable hepatocellular carcinoma with use of 90Y microspheres (TheraSphere): safety, tumor response, and survival. J Vasc Interv Radiol. 2005 Dec;16(12):1627-39. doi: 10.1097/01.RVI.0000184594.01661.81. PMID 16371529
- [Background] Vente MA, Wondergem M, van der Tweel I, van den Bosch MA, Zonnenberg BA, Lam MG, van Het Schip AD, Nijsen JF. Yttrium-90 microsphere radioembolization for the treatment of liver malignancies: a structured meta-analysis. Eur Radiol. 2009 Apr;19(4):951-9. doi: 10.1007/s00330-008-1211-7. Epub 2008 Nov 7. PMID 18989675
- [Background] Dawson LA, Guha C. Hepatocellular carcinoma: radiation therapy. Cancer J. 2008 Mar-Apr;14(2):111-6. doi: 10.1097/PPO.0b013e31816a0e80. PMID 18391616
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Background] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Background] Kulik LM, Carr BI, Mulcahy MF, Lewandowski RJ, Atassi B, Ryu RK, Sato KT, Benson A 3rd, Nemcek AA Jr, Gates VL, Abecassis M, Omary RA, Salem R. Safety and efficacy of 90Y radiotherapy for hepatocellular carcinoma with and without portal vein thrombosis. Hepatology. 2008 Jan;47(1):71-81. doi: 10.1002/hep.21980. PMID 18027884
- [Derived] Mazzaferro V, Sposito C, Bhoori S, Romito R, Chiesa C, Morosi C, Maccauro M, Marchiano A, Bongini M, Lanocita R, Civelli E, Bombardieri E, Camerini T, Spreafico C. Yttrium-90 radioembolization for intermediate-advanced hepatocellular carcinoma: a phase 2 study. Hepatology. 2013 May;57(5):1826-37. doi: 10.1002/hep.26014. Epub 2013 Mar 22. PMID 22911442